CLINICAL TRIAL: NCT04420117
Title: Perioperative Assessment of Physical Capacity in Elderly Patients Undergoing Laparoscopic Colorectal Surgery- Atlas Study
Brief Title: Perioperative Assessment of Physical Capacity in Elderly Patients Undergoing Laparoscopic Colorectal Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Principal investigator, Hospital Universitario La Fe
Other Study IDs: Atlas
Record Dates: First submitted 2020-05-22; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Perioperative assessment of physical capacity — Evaluation of physical capacity with the Short Physical Performance Battery (SPPB) questionaire

SUMMARY:
Evaluation of preoperative physical capacity and its evolution in the postoperative period in older patients after undergoing laparoscopic surgery for colorectal cancer, with the test:

- Short Physical Performance Battery (SPPB)

After the inclusion of the first 10 patients, a preliminary feasibility study will be carried out and thus we have coverage of this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥65 years.
* ASA I-III
* Patients with absence of cognitive deficit.
* Informed consent signed prior to surgery.

Exclusion Criteria:

* Refusal of the patient to participate in the study.
* Patients with disabilities to give their consent.
* ASA IV-V.
* Pregnancy or lactation.
* Health status that prevent physical exercise, such as unstable heart disease, severe systematic disease, or serious orthopedic conditions

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing laparoscopic colorectal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the physical capacity | 21 days before surgery
  Evaluation of the physical capacity only with the Short Physical Performance Battery (SPPB) questionnaire
Evaluation of the physical capacity | 21 days after surgery
  Evaluation of the physical capacity only with the Short Physical Performance